CLINICAL TRIAL: NCT04710836
Title: The Nottingham Recovery From COVID-19 Research Platform Assessment Clinic
Brief Title: NoRCoRP Assessment Clinic
Acronym: NoRCoRP
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20RM056
Record Dates: First submitted 2020-12-10; First posted 2021-01-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood will be stored for later analysis of DNA. This will only be stored with the specific consent of the patient as outlined in the consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main overarching aim of this study is to build a research clinic, as part of the NoRCoRP platform covering Nottingham and Nottinghamshire to facilitate learning and research in the whole population of patients who have had COVID-19.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2 / COVID-19) pandemic, has affected over 13 million people, and caused significant worldwide mortality and morbidity. Frequent long-term respiratory complications include persistent breathlessness and fatigue, with potential for ongoing organising pneumonia and new pulmonary fibrosis as well as thromboembolic disease. Additional features seen in at least some patients post hospital include impaired musculoskeletal function, impaired renal function, neurological impairment, cardiac dysfunction and significant psychiatric morbidity.

The majority of patients with COVID-19 were not admitted to hospital, and the longer-term consequences of infection with SARS-CoV-2 in this much larger patient group are unknown. Whilst many patients had relatively mild disease and made a good recovery, a significant number have been left with symptoms similar to those who were admitted to hospital.

In setting up a post COVID-19 respiratory review clinic, we expect to generate new findings, support studies that have already been submitted for funding, to provide a focus for further grant funding, and to provide an infrastructure to support new clinical trials. We also expect the insights gained from research using this platform to be of value for service planning in the region and beyond. We will prioritise patients who were not admitted to hospital but who have been left with significant morbidity by establishing this new General Practitioner (GP) referral research clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) referred into the post COVID-19 respiratory outpatient clinic from primary care, following a swab, imaging or strong clinical diagnosis of COVID-19
* Adults discharged from hospital with a clinical diagnosis of COVID-19 (who are not included in the PHOSP-COVID study)

Exclusion Criteria:

* Children (<18 years) referred into the post COVID-19 respiratory outpatient clinic. This clinic is only open to adults and referrals for children will not be accepted
* Adults discharged from hospital with a clinical diagnosis of COVID-19 and have been included in the PHOSP-COVID study
* Patients unable to provide informed consent by themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have previous had a diagnosis of COVID-19 and have been referred into a post-COVID-19 respiratory outpatients clinic from primary care due to ongoing complications related to the COVID-19 diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with symptoms at presentation to the research clinic | September 2020 - August 2024
  Patient reported symptoms
Short Physical Performance Battery | September 2020 - August 2024
  Assessment of functional capacity
Quadricep muscle strength | September 2020 - August 2024
  Assessment of functional capacity using a handheld dynamometer
Chalder's Fatigue Score | September 2020 - August 2024
  Assessment of fatigue using the Chalder 11-item fatigue questionnaire
Number of participants with rehabilitation needs at presentation to clinic | September 2020 - August 2024
  Rehabilitation needs based on clinical assessment by a multidisciplinary team (musculoskeletal, cognitive and cardiopulmonary)
EQ-5D-5L | September 2020 - August 2024
  Assessment of generic health status using the EQ-5D-5L questionnaire
Montreal Cognitive Assessment | September 2020 - August 2024
  Assessment of cognitive state using the MoCA questionnaire

SECONDARY OUTCOMES:
Anxiety and Depression | September 2020 - August 2024
  Derived by completion of the Hospital Anxiety and Depression Scale (HADS) questionnaire
Pittsburgh Sleep Quality Index | September 2020 - August 2024
  Assessment of sleep quality using the PSQI questionnaire
Healthcare service needs following COVID-19 diagnosis | September 2020 - August 2032
  Monitoring of NHS records for incidence of re-presentation to primary or secondary care related to COVID-19 complications and survival.
Biological markers of recovery from COVID-19 | September 2020 - August 2032
  Assessment of blood taken for clinical purposes (where available) including renal function, liver function, full blood count, HbA1C, Brain natriuretic peptide, vitamin D, thyroid function, C-reactive protein (CRP), Creatine kinase for markers of COVID-19 recovery. Batched inflammatory and metabolic markers as well as whole blood DNA will also be assessed from stored samples.
Fried Frailty Index | September 2020 - August 2024
  Frailty assessment covering: shrinking, exhaustion, physical activity, slowness and weakness domains.
Body composition | September 2020 - August 2024
  Body composition derived from bioelectrical impedance analysis to determine: body mass index, fat free mass index, fat free mass (kg), fat mass (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bolton, Principal Investigator — University of Nottingham & Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham City Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No